CLINICAL TRIAL: NCT04301726
Title: Efficacy of Deutetrabenazine in Huntington's Disease Patients with Dysphagia: a Randomised, Placebo-controlled Pilot Study
Brief Title: Efficacy of Deutetrabenazine to Control Symptoms of Dysphagia Associated with HD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated prematurely due to the lack of availability of the study drug.
Sponsor: Fundacion Huntington Puerto Rico (Other)
Responsible Party: Principal Investigator, Sylvette Ayala-Pena, Scientific Official/Principal Investigator, Fundacion Huntington Puerto Rico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2002027824
Record Dates: First submitted 2020-02-13; First posted 2020-03-10 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — deutetrabenazine

STUDY DESIGN:
Intervention Model Description: Placebo-controlled pilot study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Deutetrabenazine (Experimental): The participants randomized to this group will receive oral deutetrabenazine for 8 weeks. Week 1: 6 mg once daily; Week 2: 6 mg twice daily (BID); Week 3: 9 mg BID; Week 4: 12 BID; Week 5: 15 mg BID; Week 6: 18 mg BID; Week 7: 21 mg BID; Week 8: 24 mg BID.
  Interventions: Drug: Deutetrabenazine Oral Tablet [Austedo]
- Placebo (Placebo Comparator): The participants randomized to this group will receive oral placebo for 8 weeks. Week 1: 6 mg once daily; Week 2: 6 mg twice daily (BID); Week 3: 9 mg BID; Week 4: 12 BID; Week 5: 15 mg BID; Week 6: 18 mg BID; Week 7: 21 mg BID; Week 8: 24 mg BID.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Deutetrabenazine Oral Tablet [Austedo] — The participants randomized to this group will receive oral deutetrabenazine for 8 weeks. Week 1: 6 mg tab once daily; Week 2: 6 mg tab (BID); Week 3: 9 mg tab (BID); Week 4: 12 mg tab (BID); Week 5: 15 mg (6 mg tab + 9 mg tab BID); Week 6: 18 mg (9 mg tab + 9 mg tab BID); Week 7: 21 mg (9 mg tab + 12 mg tab BID); Week 8: 24 mg (12 mg tab BID).
  Other Names: Austedo
  Arms: Deutetrabenazine
Drug: Placebo oral tablet — The participants randomized to this group will receive oral placebo for 8 weeks. Week 1: 6 mg tab once daily; Week 2: 6 mg tab (BID); Week 3: 9 mg tab (BID); Week 4: 12 mg tab (BID); Week 5: 15 mg (6 mg tab + 9 mg tab BID); Week 6: 18 mg (9 mg tab + 9 mg tab BID); Week 7: 21 mg (9 mg tab + 12 mg tab BID); Week 8: 24 mg (12 mg tab BID).
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
To determine the efficacy of deutetrabenazine to control symptoms of dysphagia associated with HD.

DETAILED DESCRIPTION:
The primary endpoint is the change in swallow function/dysphagia from baseline to maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HD
* Symptoms of dysphagia
* Must be able to swallow tablets

Exclusion Criteria:

* Other confounding diseases that affect swallowing
* Depression
* Hepatic impairment
* Renal impairment
* Dementia

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of deutetrabenazine to control symptoms of dysphagia associated with Huntington's disease. | 18 months
  The change in swallow function/dysphagia from baseline to maintenance therapy using the clinical swallow assessment Huntington's Disease Dysphagia Scale (HDDS). The Huntington's Disease Dysphagia Scale is an 11-item scale used to monitor swallowing difficulties in persons in early to advanced disease stages. The Huntington's Disease Dysphagia Scale includes questions related to the preparatory oral, oral, pharyngeal, and esophageal phases of swallow. The response options are the following: Question 1-4 and 6-11: 1 No, almost never; 2 Yes, seldom; 3 Yes, sometimes; 4 Yes, frequently; 5 Yes, almost always. Question 5: 1 Yes, almost always; 2 Yes, frequently; 3 Yes, sometimes; 4 Yes, seldom; 5 No, almost never. Higher scores mean a worse outcome.
Non-instrumental assessment of the efficacy of deutetrabenazine to control symptoms of dysphagia associated with Huntington's disease. | 18 months
  Non-instrumental assessment and symptoms of dysphagia using the Bedside Swallowing Assessment Scale. The Bedside Swallowing Assessment Scale interpretation: Level 1: irrelevant alterations, scores ≤ 19; level 2: average alterations, scores 20-23; level 3: severe alterations, scores ≥ 24. Higher scores mean a worse outcome.
Instrumental assessment of the efficacy of deutetrabenazine to control symptoms of dysphagia associated with Huntington's disease. | 18 months
  Assessment of pharyngeal and esophageal dysphagia using the Videofluoroscopic Swallowing Study, also known as the Modified Barium Swallow Study. The instrumental assessment provides a description of any anatomical differences and physiological problems that may be associated with the patients' symptoms in all phases of the swallow. Results from the videoflourographic study are used to rate the severity of dysphagia according to the Dysphagia Outcome and Severity Scale. The Dysphagia Outcome and Severity Scale scores range from 1 to 7, with 7 representing normal swallowing and 1 representing severe dysphagia.

SECONDARY OUTCOMES:
Effect of deutetrabenazine on body weight in HD patients. | 18 months
  Secondary endpoints are treatment success from baseline to maintenance therapy on body weight. Body weight will be calculated in kilograms.
Effect of deutetrabenazine on body mass index in HD patients. | 18 months
  Secondary endpoints are treatment success from baseline to maintenance therapy on body mass index. Body mass index will be calculated by dividing the weight in kilograms by the square of the height in meters (kg/m2).
Effect of deutetrabenazine on fat distribution in HD patients. | 18 months
  Secondary endpoints are treatment success from baseline to maintenance therapy on body fat distribution. Body fat distribution will be estimated using skinfold caliper measurements of skinfold thickness at four sites: scapular, biceps, triceps and suprailiac, together with arm and leg circumferences.

OTHER OUTCOMES:
Effect of deutetrabenazine on quality of life in HD patients. | 18 months
  Treatment success from baseline to maintenance therapy on quality of life of HD patients with dysphagia. The quality of life (specifically Assessment of health status and disability using the World Health Organization Disability Assessment Schedule (WHODAS) version 2.0. The WHODAS 2.0 covers six domains of functioning including cognition, mobility, self-care, getting along, life activities and participation in community activities. The following numbers are assigned to the responses: 0= No difficulty; 1= Mild difficulty; 2= Moderate difficulty; 3= Severe difficulty; and 4= Extreme difficulty or can't do. In this test of global day-to-day functioning, higher scores indicate worse functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacion Huntington Puerto Rico, Inc. - Huntington's disease Clinic, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No